CLINICAL TRIAL: NCT05032534
Title: Examination of a New Irrigation System for Transanal Irrigation in Children With Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Qufora A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Højt skyl
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-08

CONDITIONS: Fecal Incontinence; Constipation - Functional
Keywords: Transanal irrigation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: The children will use either the old or the new cone for transanal irrigation for 6 weeks and then crossover to the contrary cone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly developed cone for 6 weeks the currently used cone for 6 weeks (Active Comparator): Starts off with treatment with the newly developed cone for transanal irrigation for 6 weeks and are then instructed to crossover to the contrary system, the currently used, for additional 6 weeks.
  Interventions: Device: Cone Small, Qufora A/S; Device: Colotip, Coloplast A/S
- Currently used cone for 6 weeks the newly developed cone for 6 weeks (Active Comparator): Starts off with treatment with the currently used cone for transanal irrigation for 6 weeks and are then instructed to crossover to the contrary system, the currently used, for additional 6 weeks.
  Interventions: Device: Cone Small, Qufora A/S; Device: Colotip, Coloplast A/S

INTERVENTIONS:
Device: Cone Small, Qufora A/S — Newly developed cone in a softer material and a design matching the use for transanal irrigation.
Device: Colotip, Coloplast A/S — Cone currently used for transanal irrigation at the Pediatric Ward, Aarhus University Hospital.

SUMMARY:
The aim of this study is to investigate if a new irrigation system for transanal irrigation (TAI) is effective and more tolerable than the currently used system at the Pediatric Ward at Aarhus University Hospital.

DETAILED DESCRIPTION:
This is a randomized, controlled study.

This study will be performed at Aarhus University Hospital (Denmark) and Aalborg University Hospital (Denmark) following the same protocol.

According to the initial randomization, children will be allocated to treatment with the new system (group A) or with the currently used system (group B). After a period of 6 weeks the child will crossover to use the contrary system.

The hypothesis is that A TAI system specifically developed for children will enhance the child's toleration of irrigation due to fewer reports on pain at insertion which will lead to better compliance. This outcome will induce a comparable or better effect on their fecal incontinence and reduce the needed follow-up period due to fewer incontinence relapse.

ELIGIBILITY:
Inclusion Criteria:

* Fecal incontinence on neurogenic or non-neurogenic basis, where transanal irrigation is indicated.

Exclusion Criteria:

* Morbus Hirschsprungs disease.
* Anorectal malformations.
* Use of medication that are known to cause constipation (e.g. anticholinergics)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The effect on fecal incontinence episode frequency | 12 weeks
  Evaluated by home recordings.
Evaluation of discomfort and on pain assessed on a Visual Analog Scale | 12 weeks
  Evaluated by home recordings.

SECONDARY OUTCOMES:
Extent of constipation | 12 weeks
  Evaluated by home recordings and transabdominal rectal ultra sound.
Evaluation of urinary incontinence episodes | 12 weeks
  Evaluated by home recordings.
Evaluation of compliance assessment using the different systems | 12 weeks
  Evaluated by home recordings.
Estimation in changes of the child's well-being | 12 weeks
  Evaluated by home recordings using WHO-5

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Aalborg University Hospital, Aalborg, The North Denmark Region

IPD SHARING:
Plan to Share IPD: Undecided